CLINICAL TRIAL: NCT02985281
Title: Safety and Efficacy of Gratisovir (Sofosbuvir)- Ribavirin Daul Therapy in Egyptian Pediatric Patients With Chronic Hepatitis C Infection. A Prospective, Randomized, Multicenter Study
Brief Title: Safety and Efficacy of Gratisovir (Sofosbuvir)- Ribavirin Therapy in Pediatric Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Liver Institute, Egypt (Other)
Collaborators: Pharco Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Samira Abdel-Wahab Abdel- Aziz, lecturer of pediatric hepatology., National Liver Institute, Egypt
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 00114/2016
Record Dates: First submitted 2016-11-21; First posted 2016-12-07 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Pharmacological Action
Keywords: direct acting antiviral drugs, chronic hepatitis C virus infection
MeSH Terms: interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): 20 patients will be randomly assigned into arm 1; treated for fixed 24 duration with Gratisovir (Sofosbuvir) and Ribavirin. First intervention 'Sofosbuvir oral product' 200 mg tablet with food on daily doses based on body weight (20-29.9 kg will take one 200 mg tab daily); (30-39.9 kg will take 1.5 tab 200 mg daily); (> 40 kg will take 2 tab 200 mg daily).
  Second intervention 'Ribavirin oral product' 200 mg tab on (15 mg/kg daily) doses based on body weight.
  Interventions: Drug: Sofosbuvir Oral Product; Drug: Ribavirin
- Arm 2 (Active Comparator): 20 patients will be randomly assigned into arm 2; treated as response guided duration; patient who show very rapid virological (undetectable HCV RNA after 2 weeks) will be treated for 16 weeks duration and reset will complete the 24 weeks duration.
  Intervention 'Sofosbuvir Oral Product' 200 mg tablet with food on daily doses based on body weight (20-29.9 kg will take one 200 mg tab daily); (30-39.9 kg will take 1.5 tab 200 mg daily); (> 40 kg will take 2 tab 200 mg daily).
  Second intervention 'Ribavirin oral product' 200 mg tab on (15 mg/kg daily) doses based on body weight.
  Interventions: Drug: Sofosbuvir Oral Product; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir Oral Product — direct acting antiviral drug for HCV infection
  Other Names: Gratisovir
Drug: Ribavirin — antiviral drug for HCV infection

SUMMARY:
Evaluation of Safety and Efficacy of Gratisovir (Sofosbuvir)- Ribavirin Therapy in Egyptian Pediatric Patients With Chronic Hepatitis C Infection aged 10- 18 years old.

DETAILED DESCRIPTION:
Male or female child ≥ 10 years and ≤ 18 years of age chronically infected with hepatitis C virus, willing and able to complete all study visits and procedures. Acceptance from the parents will be recruited for giving a verbal and written informed consent. Patient with childs Pugh class B or C, compensated cirrhosis may be enrolled. Patient with cirrhosis with their alpha fetoprotein is more than 100 ng/ml and patient with coinfection of Hepatitis B virus or HIV will be excluded. Participation in the study procedures is anticipated to last up to 40 weeks including a screening and eligibility assessment phase (4 weeks duration), a 24- week treatment phase, and 12- week post treatment follow up phase.

A detailed treatment log of the returned investigational product will be established with the investigator (or the pharmacist) and countersigned by the investigator and the monitoring team.

Compliance is assessed by counting the number of returned tablets at each visit.

A discontinuation is defined as a period with at least seven consecutive days without study drug intake.

Safety and efficacy will be compared between cirrhotic versus non-cirrhotic subjects in multivariate model to test the impact of this pretreatment characteristic on safety, tolerability and efficacy endpoints.

Safety analysis:clinical adverse events will be displayed by body system (soc) for each study subject and by treatment group, using MedDRA coding. Summary of statistics of safety and efficacy endpoints will be displayed by stratification parameters.

ELIGIBILITY:
Inclusion Criteria:

Male or female child ≥ 10 years and ≤ 18 years of age chronically infected with hepatitis C virus.

willing and able to complete all study visits and procedures. Acceptance from the parents will be recruited for giving a verbal and written informed consent.

Patient with child,s Pugh class B or C, compensated cirrhosis may be enrolled.

Exclusion Criteria:

1. Patient with cirrhosis with their alpha fetoprotein is more than 100 ng/ml.
2. Patient with coinfection of hepatitis B virus or Human Immunodeficiency Virus will be excluded.
3. Creatinine clearance < 50 ml/minute.
4. Albumin<3 gm/dl.
5. aspartate aminotransferase or alanine aminotransferase > 10 upper limit of normal.
6. Pregnant and lactating females.
7. Associated morbidity such as uncontrolled diabetes mellitus, schistosomiasis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of SVR12 in both treatment groups after 12 following completion of treatment (SVR12) | 40 weeks including a screening and eligibility assessment phase (4 weeks duration), a 24- week treatment phase, and 12- week post treatment follow up phase.
  incidence of SVR12 in both treatment groups after 12 weeks following completion of treatment (SVR12)

SECONDARY OUTCOMES:
assessment of the nature, severity and frequency of the adverse effects and absolute values and changes over time from pre-dose values for hematology clinical chemistry, urine analysis, vital signs and ECG parameters. | 40 weeks including a screening and eligibility assessment phase (4 weeks duration), a 24- week treatment phase, and 12- week post treatment follow up phase.
  Safety and tolerability are assessed by: the nature, severity and frequency of the adverse effects and absolute values and changes over time from pre-dose values for hematology clinical chemistry, urine analysis, vital signs and ECG parameters. Clinical adverse events will be displayed by body system (SOC) for each study subject and by treatment group, using MedDRA coding. Absolute laboratory values, changes and its graded abnormalities will be displayed) for each study subject and by treatment group. The proportions of subjects experiencing Clinical adverse events and laboratory abnormalities of a given type will be computed and presented along with descriptive statistics. Vital signs data will be similarly assessed, and any post baseline changes in physical examination findings will be summarized in tubular form, by subject and by treatment cohort.
  Summary statistics of efficacy and safety end points will be displayed by stratification parameters

CONTACTS AND LOCATIONS:
Overall Officials: Behairy Behairy, professor, Study Director — National Liver Institute, Egypt
Locations (1):
- National liver institute, Sijīn al Kawm, Menofia, Egypt

IPD SHARING:
Plan to Share IPD: No